CLINICAL TRIAL: NCT05856344
Title: A Study for Crossability of Novel Spherical Tip Versus Regular Noncompliant Balloon in Tortuous Coronary Artery Postdilatation：A Multicenter, Randomized, Controlled, Single Blind Trial
Brief Title: A Study for Crossability of Spherical Tip Versus Regular Noncompliant Balloon in Tortuous Coronary Artery Postdilatation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Hospital of China Medical University (Other)
Collaborators: The People's Hospital of Liaoning Province (Other)
Responsible Party: Principal Investigator, Yingxian Sun, Chief of Department of Cardiology in First Hospital of China Medical University, First Hospital of China Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: [2023]25
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Spherical Tip; Noncompliant Balloon; Postdilation; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spherical tip noncompliant balloon (Experimental): Enrolled patients who were randomly assigned to this group underwent stent postdilation using the spherical tip non compliant balloon(APT Medical Inc，CONQUEROR NC Pro). The selection of balloon size is based on the expected target lesion stent diameter, and the length range is restricted among 8-12mm. It will be defined as balloon passage failure if it fails to pass the target lesion after three attempts. After that, based on the purpose of completing the surgery, alternative options can be selected based on the surgeon's experience, including double-guide wire assistance, 5in6 support, the use of regular noncompliant balloon and so on.
  Interventions: Device: Spherical tip noncompliant balloon
- Regular noncompliant balloon (Active Comparator): Enrolled patients who were randomly assigned to this group underwent stent postdilation using the regular noncompliant balloon(tapered-tip). The selection of balloon size is also based on the expected target lesion stent diameter, and the length range is restricted among 8-12mm. It will be defined as balloon passage failure if it fails to pass the target lesion after three attempts. After that, based on the purpose of completing the surgery, alternative options can be selected based on the surgeon's experience, including tip modification, double-guide wire assistance, 5in6 support, the use of spherical tip non compliant balloon(APT Medical Inc，CONQUEROR NC Pro) and so on.
  Interventions: Device: Regular noncompliant balloon

INTERVENTIONS:
Device: Spherical tip noncompliant balloon — The main difference of this experimental balloon is the spherical tip, other parameters are consistent with regular noncompliant balloons.
  Arms: Spherical tip noncompliant balloon
Device: Regular noncompliant balloon — The balloon is designed as tapered-tip.
  Arms: Regular noncompliant balloon

SUMMARY:
The goal of this clinical trial is to compare the crossability of novel spherical tip versus regular noncompliant balloon in CHD population with tortuous coronary artery leisions that requiring postdilation after stent implantation.

The main question it aims to answer is:

•Wether the spherical tip balloon have advantages in terms of crossability compared to regular noncompliant balloons Participants will sign an informed consent form, collaborate with data collection, and accept the intervention measures from corresponding groups. Researchers will compare spherical tip balloon with regular noncompliant balloon to see if there is any difference in crossability.

DETAILED DESCRIPTION:
The tortuous lesion increases the difficulty of coronary intervention treatment, especially when there is still a large angle after stent implantation. The ability of the non compliant balloon to pass through the stent segment becomes the key to complete the operation.

The spherical tip noncompliant balloon is an original design by our center, which reduces its resistance to stent struts through the spherical structure of balloon tip, and is committed to increasing the crossability of the balloon.This study is a multicenter, randomized, single blind design with the aim of truly revealing the differences in parameters such as success rate of crossing, times of attemptation, and time consumption between the novel spherical tip and regular non compliant balloon.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old, regardless of gender
* Patients with indications for coronary artery stent implantation
* The vascular curvature angle<120 ° after coronary artery stent implantation
* Noncompliant balloon postdilation is required
* Voluntarily participate and sign an informed consent form

Exclusion Criteria:

* Pregnant women or patients who are attempting to get pregnant
* Patients participating in clinical trials of other drugs or medical devices
* Patients deemed unsuitable by the researchers to participate in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Success passage rate at the first attempt | From start to end of surgery
  The success passage rate of the noncompliant balloon through the tortuous target lesion at the first attempt

SECONDARY OUTCOMES:
The final success passage rate | From start to end of surgery
  The final success passage rate of the noncompliant balloon through the tortuous target lesion under three attempts
The number of attempts | From start to end of surgery
  The number of attempts required for the noncompliant balloon to pass through the tortuous target lesion
The time required | From start to end of surgery
  The time required for the noncompliant balloon to pass through the tortuous target lesion
Major adverse cardiac event | 3 months after percutaneous coronary intervention
  defined as death from all, cardiac, or noncardiac causes, myocardial infarction, repeat revascularization and stroke during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Yingxian Sun, Phd, Principal Investigator — First Hospital of China Medical University
Locations (1):
- First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided